CLINICAL TRIAL: NCT00300599
Title: A Randomized Controlled Study of the Long-term Effects of Nasal Continuous Positive Airway Pressure on Systemic Blood Pressure, Coagulability and Carotid Intima-media Thickness in Obstructive Sleep Apnea Syndrome
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) on Systemic Blood Pressure, Coagulability and Carotid Intima-media Thickness in Patients With Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resp/hui/2006/001
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Continue positive airway pressure
  Interventions: Device: Continuous Positive Airway pressure
- B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Continuous Positive Airway pressure — Continuous positive pressure device with a time clock
  Arms: A
Other: Placebo — Placebo
  Arms: B

SUMMARY:
Sleep-disordered breathing (SDB) briefly means cessation of breathing during sleep at least 5 times per hour. Sleep-disordered breathing affects 9 to 24% of the middle-aged and overall 4% of the middle-aged males suffers from Obstructive sleep apnea syndrome (OSAS) i.e. SDB with associated daytime sleepiness. Several major epidemiological studies have shown that SDB is not only an independent risk factor for systemic hypertension but it is also associated with cardiovascular complications such as heart failure, stroke, and sudden death.

The mechanisms for the linkage between Sleep-disordered breathing and cardiovascular diseases are not fully determined but surges in sympathetic nerve activity are seen at the end of each apneic episode accompanied by large rises in systemic arterial blood pressure (BP). The increased levels of muscle sympathetic nerve activity are diminished by nasal continuous positive airway pressure (CPAP) therapy. Numerous studies have found a hypercoagulable state in terms of increased clotting factor and platelet activities, and impaired fibrinolysis in coronary artery disease, ischaemic stroke, and sleep-disordered breathing. Common carotid artery intima-media thickness (IMT) has been shown to correlate with traditional vascular risk factors and may predict the likelihood of acute coronary events and stroke. Recently, carotid artery intima-media thickness has been shown to have positive correlations with the severity of sleep disordered breathing.

Despite robust evidence showing improvement of symptoms, cognitive function and quality of life in patients with obstructive sleep apnea treated with nasal continuous positive airway pressure, there are conflicting short-term data whether continuous positive airway pressure can reduce blood pressure in patients with obstructive sleep apnea. This randomized controlled study aims to assess the long-term effects of nasal continuous positive airway pressure on 1) 24 hr systemic blood pressure; 2) Coagulation state; and 3) Carotid artery intimal media thickness.

DETAILED DESCRIPTION:
Subjects and Methods: We propose to carry out a prospective, randomized controlled study on 100 consecutive patients newly diagnosed with obstructive sleep apnea syndrome, as defined by overnight sleep study showing Apnea- hypopnoea index (AHI) >or=5 per hour of sleep plus Epworth sleepiness scale (ESS) ≥10.1 The patients will be recruited from the Respiratory Clinic, Prince of Wales Hospital (PWH), Shatin.

Sleep assessment: Overnight diagnostic polysomnography(PSG) [Healthdyne Alice 4, USA] will be performed at Prince of Wales Hospital, Hong Kong for every subject on the first night recording electroencephalogram, electro-oculogram, submental electromyogram, bilateral anterior tibial electromyogram, electrocardiogram, chest and abdominal wall movement by inductance plethysmography, airflow measured by a nasal pressure transducer [PTAF2, Pro-Tech, Woodinville, WA, USA]and supplemented by oronasal airflow thermister, and finger pulse oximetry as in our previous studies.2,3 Sleep stages will be scored according to standard criteria by Rechtshaffen and Kales.4 Apnoea is defined as cessation of airflow for > 10 seconds and hypopnea as a reduction of airflow of > 50% for > 10 seconds plus an oxygen desaturation of > 3% or an arousal.

Ambulatory Blood Pressure Monitoring (ABPM):

All patients with obstructive sleep apnea syndrome will be fitted with the Ultralite Ambulatory Blood Pressure Monitoring (Spacelabs Medical, Redmond, WA) via an arm cuff as out-patients during normal activities and monitored for 48 hrs prior to commencement of continuous positive airway pressure or conservative treatment. The patients' arm circumference will be measured at the biceps level and an appropriate sized arm cuff will be applied. The machine will be programmed for cuff inflation measurement every 30 minutes for 48 hrs and can only be removed for bathing. Patients will be asked to abstain from caffeine-containing products during this time but to continue their normal daily activities. Patients will record the time they retire to bed and the subsequent time of waking in order to identify the sleep period. Data gathered before 6pm on the second evening will be discarded to allow for acclimatization and the analysis will be performed with the second 24 hr of data (6pm to 6am).5 Data will be manually checked for artifact by our respiratory fellow, who will be blinded to the treatment status of the patient. Ambulatory Blood Pressure Monitoring will be repeated for all patients with significant OSAS at 3, 6, and 12 months of the study.

Conservative treatment 6 months followed by continuous positive airway pressure 6 months vs Concurrent continuous positive airway pressure+ Conservative treatment for 12 months:

Following confirmation of significant obstructive sleep apnea syndrome from the overnight sleep study with Apnoea hyponea index ≥ 5/hr and Epworth Sleepiness Scale ≥10 and completion of baseline Ambulatory Blood Pressure Monitoring, each patient will be interviewed by the physician on duty and randomized by computer into either Group 1) Conservative treatment for the first 6 months followed by therapeutic Continuous positive airway pressure for the next 6 months or Group 2) Conservative treatment plus therapeutic Continuous positive airway pressure for 12 months. As sleepiness is the main indication for Continuous positive airway pressure treatment, we have decided that a randomized placebo controlled design is not feasible for this long-term study. The research nurse responsible for randomization of patients to different treatment arms will not participate in outcome assessments, which will be conducted by a different team of nurses who are not aware of the randomization status of the patients.6,7 Group 1: After confirmation of significant obstructive sleep apnea syndrome, the patients will be informed about the nature of their disease and the need to start treatment. They are encouraged to a) avoid sleep deprivation by having sufficient hours of sleep every night; b) sleep in lateral positions; c) avoid sedatives and alcohol consumption; and d) lose weight by following a home diet prescribed by a dietitian.8 The patients will be reviewed at the respiratory clinic at 1, 3 and 6 months to re-assess their sleepiness & body mass index. Ambulatory blood pressure monitoring will be repeated at 3, 6, and 12 months. On completion of the conservative treatment and evaluation including ambulatory blood pressure monitoring at 6 months, patients in group 1 will be started on therapeutic continuous positive airway pressure treatment, as outlined under group 2, after an overnight continuous positive airway pressure titration study.

Group 2: Patients in the therapeutic continuous positive airway pressure arm will be given a short trial of continuous positive airway pressure therapy with the Autoset (Resmed, Sydney, Australia) device for approximately 30 minutes for acclimatization in the afternoon. Each patient will be given a basic CPAP education programme by our respiratory nurse supplemented by education brochure.2 Attended continuous positive airway pressure titration will be performed with the Autoset auto-titrating device on the second night of the polysomonograph study. All patients will be prescribed the Horizon LT 8001 continuous positive airway pressure device (De Vilbiss, Somerset, PA, USA) with a time counter recording machine run time. The continuous positive airway pressure pressure for each patient will be set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night as determined by the overnight Autoset continuous positive airway pressure titration study. 2,3 The patients will be followed up at the Respiratory clinic at 1, 3, 6, and 12 months and the objective continuous positive airway pressure compliance will be measured from the time counter. All patients in each arm will be followed up at the Respiratory clinic regularly and the objective continuous positive airway pressure usage will be measured from the time counter.

Other outcome assessment:

Prior to commencement of conservative treatment or nasal continuous positive airway pressure , all patients have to go through several measurements. These include assessment of subjective sleepiness with the Epworth sleepiness scale (ESS),9 quality of life with the Calgary Sleep Apnoea Quality of Life Index (SAQLI), 10 hemostatic assays (DD, TAT, fibrinogen, vWF:ag),11 and evaluation of carotid artery initimal media thickness.12-14 The ESS is a questionnaire specific to symptoms of daytime sleepiness and the patients are asked to score the likelihood of falling asleep in eight different situations with different levels of stimulation, adding up to a total score of 0 to 24.9 The Calgary Sleep Apnea Quality of Life Index (SAQLI) has 35 questions organized into four domains: daily functioning, social interactions, emotional functioning and symptoms with a fifth domain, treatment-related symptoms, to record the possible negative impacts of treatment. It contains items shown to be important to patients with sleep apnea and is designed as a measure of outcome in clinical trials in sleep apnea.10 The early version of the Calgary Sleep Apnea Quality of Life Index (SAQLI) was applied previously to our study on Chinese obstructive sleep aonoea patients on continuous positive airway pressure 2 but an updated version will be applied to this study.15 Carotid artery intimal media thickness will be assessed with B-mode Doppler according to a standardized scanning protocol for the right and left carotid arteries using images of the far wall of the distal 10 mm of the common carotid arteries as described by Woo et al previously.12-14 Carotid scans will be analyzed with a computerized edge-detection system that have previously been described and validated.12,16 Two end-diastolic frames are selected, digitized, and analyzed for mean intimal media thickness, and the average reading from these 2 frames is calculated for both right and left carotid arteries. The carotid scan operator is blinded to the identity of studied subjects and stage of the study.

Hemostatic assays: After resting for 20 min in the sitting position, blood is obtained following the polysomongraphy recording through an indwelling 22-gauge venous forearm cannula that has been inserted the night before to minimize hemostatic activation due to emotions related to an impending venepuncture.11 The first 2 ml of blood will be discarded and another 15 ml of blood will be drawn into sterile ethylenediamine-tetra acetic acid (EDTA)- containing tubes (Becton Dickinson Vacutainer Systems; Franklin Lakes, New Jersey, USA). Plasma samples are obtained by centrifugation in plastic tubes at -80C until further processing. Plasma TAT and DD levels are measured by ELIZA as per the manufacturers instructions (Enzyme Research Laboratories Inc., South Bend, Indiana, USA and Diagnostica Stago, Asnieres, France). Plasma fibrinogen levels (g/l) are determined using a commercially available assay (Thrombo-S, Dade Behring, Germany). Plasma levels of vWF:ag are measured following a previously described ELISA 17 using commercial antibodies (DAKO Corp., Carpinteria, California, USA) and substrate (Bio-Rad Laboratories, Hercules, California, USA).

Primary outcome of interest: Changes in mean systemic blood pressure between group 1 and group 2 at 6 months.

Secondary outcome of interest: Changes in systolic and diastolic blood pressure between the 2 groups at 6 & 12 months; serial changes of carotid intimal media thickness between the two treatment groups over 12 months; serial changes in hemostatic assays (TAT, DD, fibrinogen, vWF:ag) between the two groups at 1 month and 6 months after treatment; Continuous positive airway pressure compliance at 6, and 12 months; Epworth Sleepiness Scale (ESS) and the Calgary Sleep Apnea Quality of Life Index (SAQLI) at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 yrs
* Apnoea Hypopnea index ≥5/hr on Polysomnography with Epworth Sleepiness Scale ≥10

Exclusion Criteria:

* Predominantly central sleep apnoea
* Recent myocardial infarction 3 months before the study
* Unstable angina
* Underlying malignancy
* Professional drivers and those handling dangerous machinery
* Patients will be considered dropouts if anti-hypertensive medication is accidentally changed by the patients or their general practitioners

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2018-02-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure measurement | 6 and 12 months

SECONDARY OUTCOMES:
Changes in systolic and diastolic Blood pressure between the 2 groups at 6 & 12 months | 6 and 12 months
serial changes of carotid intimal media thickness between the two treatment groups over 12 months | 12 months
serial changes in haemostatic assays | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, New Territories, Hong Kong